CLINICAL TRIAL: NCT02724839
Title: Innovations in the Management of Obesity and Inactivity in Pediatric Primary Care
Brief Title: Supporting Together Exercise and Play and Improving Nutrition
Acronym: STEP IN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-3406
Record Dates: First submitted 2016-03-14; First posted 2016-03-31 (Estimated); Results first posted 2020-11-03 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2019-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Biweekly Arm (Experimental): 6 group nutrition sessions co-led by a peer and a content expert, Fitbit given to parent-child dyads during second session. Sessions took place biweekly.
  Interventions: Behavioral: Group nutrition sessions; Device: Fitbit
- Monthly Arm (Experimental): 6 group nutrition sessions co-led by a peer and a content expert, Fitbit given to parent-child dyads during second session. Sessions took place monthly.
  Interventions: Behavioral: Group nutrition sessions; Device: Fitbit
- Weekly (Experimental): 6 group nutrition sessions co-led by a peer and a content expert, Fitbit given to parent-child dyads during second session. Sessions took place weekly.
  Interventions: Behavioral: Group nutrition sessions; Device: Fitbit

INTERVENTIONS:
Behavioral: Group nutrition sessions — The intervention will consist of 6 nutrition group sessions co-led by parent and a professional from the community who will rotate at each session. Group nutrition sessions will consist of a facilitated discussion of benefits and barriers to healthy eating, a short lesson led by the content expert, and a fun game or activity to reinforce the lesson. Three non-concurrent phases of the study will compare the efficacy of the group sessions when offered biweekly (Arm 1), monthly (Arm 2) and weekly (Arm 3).
  Other Names: Peer-led Group Sessions
Device: Fitbit — Parent and child dyads will each receive a Fitbit Flex wearable device at the second session. This device will be used by participants and investigators to motivate and track participants' physical activity for up to 9 months.

SUMMARY:
The purpose of this study is to design, pilot, and tweak a series of peer-led group nutrition sessions for primary care patients aged 6 -12 years who are overweight or obese and who want to eat healthier and be more active.

DETAILED DESCRIPTION:
In addition to the group nutrition sessions, the investigators will give a Fitbit to each of a parent and child dyad, which will be used to track and motivate their activity. The investigators hypothesize an improvement pre-post in children's physical activity levels, self-efficacy and intentions for physical activity, self-reported consumption of fruits, vegetables, and child quality of life, and a decrease in consumption of sugar-sweetened beverages and fast and snack-food, and television (TV)/ videos screen time

ELIGIBILITY:
Inclusion Criteria:

* Patients whose primary medical home is the Pediatric Primary Care Center (primarily Medicaid or self-pay)
* BMI is greater than 85th%ile for age and sex
* English speaking
* have access to a computer/internet or a smart phone (for uploading Fitbit data)

Exclusion Criteria:

* Have been seen in a weight management clinic within the last 2 years
* prescribed an atypical antipsychotic
* non-ambulatory

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Copeland, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Pediatric Primary Care Center (PPC) Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This was a small, iterative feasibility study as a precursor to a larger clinical trial.

REFERENCES:
- [Background] Saunders RP, Pate RR, Felton G, Dowda M, Weinrich MC, Ward DS, Parsons MA, Baranowski T. Development of questionnaires to measure psychosocial influences on children's physical activity. Prev Med. 1997 Mar-Apr;26(2):241-7. doi: 10.1006/pmed.1996.0134. PMID 9085394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 36 parent-child dyads (72 individual participants) were consented and enrolled over the entire course of the study starting with recruitment in February 2016 and ending with the final session in July 2018.
Groups:
- Biweekly Arm: 13 parent-child dyads were enrolled in this arm which convened biweekly.
- Monthly Arm: 12 parent-child dyads were enrolled in this arm which convened monthly.
- Weekly Arm: 8 parent-child dyads were enrolled in this arm which convened weekly.
Period: Overall Study
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Started | 13 | 12 | 11
Completed | 12 | 8 | 6
Not Completed | 1 | 4 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 3 | 2
Not completed — Physician Decision | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Biweekly Arm: The intervention consisted of 6 nutrition group sessions co-led by parent and a professional from the community who rotated at each session. Group nutrition sessions consisted of a facilitated discussion of benefits and barriers to healthy eating, a short lesson led by the content expert, and a fun game or activity to reinforce the lesson. This is the first of three non-concurrent phases of the study which sought to compare the feasibility and efficacy of the group sessions when offered biweekly (first phase).Parent and child dyads in each arm and phase received a Fitbit Flex wearable device at the second session.
- Monthly Arm: The intervention consisted of 6 nutrition group sessions co-led by parent and a professional from the community who rotated at each session. Group nutrition sessions consisted of a facilitated discussion of benefits and barriers to healthy eating, a short lesson led by the content expert, and a fun game or activity to reinforce the lesson. This is the second of three non-concurrent phases of the study which sought to compare the feasibility and efficacy of the group sessions when offered monthly (second phase). Parent and child dyads in each arm and phase received a Fitbit Flex wearable device at the second session.
- Weekly Arm: The intervention consisted of 6 nutrition group sessions co-led by parent and a professional from the community who rotated at each session. Group nutrition sessions consisted of a facilitated discussion of benefits and barriers to healthy eating, a short lesson led by the content expert, and a fun game or activity to reinforce the lesson. This is the third of three non-concurrent phases of the study which sought to compare the feasibility of the group sessions when offered weekly (third phase). For phases one and two participants will participate in only one phase. Due to recruitment issues in the third phase, researchers obtained IRB approval to allow participants from previous phases to participate and instead evaluated feasibility outcomes. Parent and child dyads in each arm and phase received a Fitbit Flex wearable device at the second session.
- Total: Total of all reporting groups
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm | Total
Number analyzed (Participants) | 12 | 8 | 6 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 8 | 6 | 26
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10 (2) | 8 (2) | 11 (2) | 10 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 6 | 24
  Male | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 6 | 3 | 19
  White | 1 | 1 | 3 | 5
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 8 | 6 | 26

OUTCOME MEASURES:

1. Primary Outcome: Attendance
Description: Evaluation of participant attendance in each arm.
Time Frame: Baseline, 3 months
Measure: Count of Participants; unit: Participants
Groups:
- Biweekly Arm: 12 parent-child dyads participated in the biweekly arm which convened for 6 sessions.
- Monthly Arm: 8 parent-child dyads participated in the monthly arm which convened for 6 sessions.
- Weekly Arm: 6 parent-child dyads participated in the weekly arm which convened for 6 sessions.
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 12 | 8 | 6
Participants
  Number of Participants in Attendance at Session 1 | 11 | 8 | 2
  Number of Participants in Attendance at Session 2 | 12 | 8 | 2
  Number of Participants in Attendance at Session 3 | 8 | 7 | 3
  Number of Participants in Attendance at Session 4 | 10 | 4 | 6
  Number of Participants in Attendance at Session 5 | 11 | 6 | 4
  Number of Participants in Attendance at Session 6 | 8 | 5 | 6

2. Primary Outcome: Overall Satisfaction With Group Nutrition Sessions
Description: Participants evaluated their satisfaction with the group sessions using a 5 point scale with a score of 1 being complete dissatisfaction and 5 being the greatest satisfaction.
Time Frame: Baseline, 3 months
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Biweekly Arm: 12 parent-child dyads participated in this arm which convened for 6 sessions.
- Monthly Arm: 8 parent-child dyads participated in this arm which convened for 6 sessions.
- Weekly Arm: 6 parent-child dyads participated in this arm which convened for 6 sessions.
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 12 | 8 | 6
score on a scale | 4.82 [4 to 5] | 4.68 [4 to 5] | 4.79 [4 to 5]

3. Primary Outcome: Change From Baseline in Parent-report Child's Daily Servings of Fruits and Vegetables and Time Spent on Screens.
Description: Data were not collected on any participants because we changed the study design based on qualitative participant feedback in pilot phases. Our asking participants about their habits, and showing them their data, was part of the intervention instead of an outcome to assess efficacy of the intervention.
Time Frame: Baseline, 3 months
Population: Data were not collected on any participants because we changed the study design based on qualitative participant feedback in pilot phases. Our asking participants about their habits, and showing them their data, was part of the intervention instead of an outcome to assess efficacy of the intervention.
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: PedsQL (Pediatric Quality of Life Inventory)
Description: Measure Description: PedsQL (Pediatric Quality of Life Inventory) is a modular instrument for measuring health-related quality of life in children and adolescents ages 2 to 18. Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better Health-Related Quality of Life.
Time Frame: Baseline, 3 months
Population: PEDS QL was only administered to the Biweekly Arm.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 12 | 0 | 0
score on a scale
  Baseline | 72 [53 to 85] |  |
  3 months | 74 [68 to 91] |  |

5. Secondary Outcome: BMI Z-Score
Description: BMI Z-scores compares child to age and sex matched peers. A z-score of 0 is the same as a 50th percentile in the reference population, a z-score of ± 1.0 plots at the 15th or 85th percentiles, respectively, and a z-score of ± 2 plots at roughly the 3rd or 97th percentiles. Negative numbers indicate values lower than the reference population whereas positive numbers indicate values higher than the reference population.
Time Frame: Baseline, 3 months
Population: Due to recruitment and retention issues, BMI Z-score was not evaluated for the weekly arm.
Measure: Mean (Standard Deviation); unit: score
Groups:
- Weekly Arm: Due to recruitment and retention issues, BMI Z-score was not evaluated for the weekly arm.
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 12 | 8 | 0
score | 1.84 (0.43) | 2.15 (0.41) |

6. Secondary Outcome: Number of Participants Reporting They Were Satisfied With the Group Nutrition Sessions (4 or 5 on 5-point Likert Scale)
Description: The description of the overall satisfaction variable is described in outcome #2 under primary outcomes.
Time Frame: baseline, 3 months
Population: The results for overall satisfaction are listed under outcome #2 under primary outcomes.
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Child Self-efficacy Related to Physical Activity
Description: Self efficacy was assessed using a validated 14-item questionnaire using a 5-point Strongly Agree/ Strongly Disagree scale. The range of values is 1 to 5, with lower values indicating higher self-efficacy
Time Frame: Baseline, 3 months
Population: This measure was administered at 3 months in biweekly arm and monthly arm, but not administered in weekly arm. All completed subjects contributed data in biweekly arm; 7 subjects contributed data for monthly arm.
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 12 | 7 | 0
score on a scale
  Baseline | 1.71 [1.26 to 2.39] | 2.07 [1.86 to 2.07] |
  3 months | 1.71 [1.18 to 2.00] | 1.43 [1.29 to 2.14] |

8. Secondary Outcome: Child Intention to be Active
Description: Child intention to be active was assessed with a 1-item questionnaire developed and validated by Saunders et al. This item uses a 5-point scale, with possible range of scores being 1 to 5. Higher scores indicate greater intention to be active.
Time Frame: baseline, 3 months
Population: as for outcome 7
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 12 | 7 | 0
score on a scale
  Baseline | 4.00 [3.00 to 5.00] | 4.00 [3.00 to 5.00] |
  3 months | 4.00 [4.00 to 5.00] | 4.50 [4.00 to 5.00] |

9. Secondary Outcome: Change From Baseline in Parent-reported Number of Hours of Screen Time Child Watches Daily
Description: as for outcome 3
Time Frame: Baseline, 3 months
Population: as for outcome 3
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Monthly Arm: 8 parent-child dyads participated in the biweekly arm which convened for 6 sessions.
- Weekly Arm: 6 parent-child dyads participated in the biweekly arm which convened for 6 sessions.
Arm/Group | Biweekly Arm | Monthly Arm | Weekly Arm
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8 | 0/6

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed. Difficulty recruiting and retaining engaged participants for collection of all desired outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT02724839/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT02724839/ICF_001.pdf